CLINICAL TRIAL: NCT02752503
Title: Open-label Trial on Therapeutic Effect and Tolerability of Nalmefene in Subjects With Alcohol Use Disorder and Comorbid Borderline Personality Disorder
Brief Title: Nalmefene in Alcohol Dependence and Borderline Personality Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Hospital Universitari General de Catalunya (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-NAL-2014-76
Record Dates: First submitted 2016-04-19; First posted 2016-04-27 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Alcohol Use Disorder; Borderline Personality Disorder
MeSH Terms: conditions — Alcoholism; Borderline Personality Disorder | interventions — nalmefene

ARMS (1):
- Nalmafene (Experimental)
  Interventions: Drug: Nalmefene

INTERVENTIONS:
Drug: Nalmefene

SUMMARY:
The objective is to study the effectiveness of Nalmefene in decreasing alcohol intake in subjects with alcohol use disorder and comorbid BPD.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol use disorder according to DSM 5
* Borderline personality disorder according to DSM 5
* CGI-BPD > 3
* Female have to use contraception

Exclusion Criteria:

* Other axis I disorders
* Severe organic disorder
* Pregnancy or breastfeeding
* Allergy to Nalmefene
* Subjects with Opioids use disorder or in treatment with opioid agonists

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Days of excessive alcohol intake | 2 months
  Excessive alcohol intake: >60 g in males; >40 g in females
Daily average intake (grams) | 2 months
  Daily average intake (grams)

SECONDARY OUTCOMES:
Borderline symptoms on the Borderline Symptom List - 23 (BSL-23) | 2 months
Global Impression of the Clinic on the Clinical Impression - BPD (GCI-BPD) | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Pascual, MD PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain